CLINICAL TRIAL: NCT02437396
Title: Novel Inflammatory Biomarkers Complement 5A and Hepcidin in Patients With Gaucher Disease (GD)
Brief Title: Oxidative Stress and Inflammatory Biomarkers in Gaucher Disease
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1305M34501
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Gaucher Disease Type I; Oxidative Stress; Inflammation
MeSH Terms: conditions — Gaucher Disease; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Treatment naive GD1: Type 1 Gaucher disease subjects who are naive to any treatment
- Treated GD1: Type 1 Gaucher disease who are stable on therapy (on the specific ERT and/or SRT and specific dose for at least 2 years)
- Healthy Volunteers (No longer recruiting): Age matched healthy controls. No new participants will be enrolled to this arm.

SUMMARY:
The objective of this study is to evaluate oxidative stress and/or inflammation in patients with Gaucher disease type I using a series of biomarkers and correlate with measurements of currently used diagnostic biomarkers.

DETAILED DESCRIPTION:
We will determine oxidative stress and/or inflammation related biomarkers in whole blood and/or plasma in adult subjects with Gaucher disease. Fifteen milliliter blood sample will be collected during three independent visits over a period of approximately 3 months. These samples will be processed to separate plasma from red blood cells and frozen until assays are performed. Standardized immunoassay methods and LC/MS based methods will be adopted to assay a series of biomarkers in these samples. These data will be correlated with currently used diagnostic biomarkers.

ELIGIBILITY:
Inclusion criteria:

1. All participants must be 18 years or older.
2. All enrollees must understand and cooperate with requirements of the study in the opinion of the investigators and must be able to provide written informed consent.
3. Individuals with Gaucher disease who are medically stable for participation in study in the opinion of the investigator.
4. GD subjects must be stable on a specific ERT and/or SRT therapy at a specific dose (for e.g. on a units/kg basis) for at least 2 years or be naïve to these therapies (no therapy for 2 years).
5. GD1 patients, who have had a change in therapy i.e. a change in dose or switch from one drug to another, can be enrolled after at least 6 months have elapsed since the change and is considered stable in the opinion of the clinician providing care to the patient.
6. All participants must not have taken antioxidants coenzyme Q-10, vitamin C, or vitamin E for 3 weeks prior to the study.

Exclusion Criteria:

1. Medically unstable conditions in any group as determined by the investigators
2. Concurrent disease; medical condition; or an extenuating circumstance that, in the opinion of the investigator, might compromise subject safety, study compliance, completion of the study, or the integrity of the data collected for the study.
3. Females who are pregnant or lactating or of child-bearing age who are not using acceptable forms of contraception
4. History of asthma that is presently being treated
5. Subjects who cannot or are unwilling to have blood drawn
6. Unable to adhere to study protocol for whatever reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 Gaucher disease subjects who are either naive to treatment or are stable on therapy (specific Enzyme Replacement Therapy (ERT) / Substrate Reduction Therapy (SRT) formulation at a specific dose) for at least 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Plasma C5a Concentration | 6 months
  Outcome will be reported as the change in plasma concentration of C5a (ng/ml) from baseline to 6 months in participants with Gaucher disease type 1
Change in Plasma Hepcidin Concentration | 6 months
  Outcome will be reported as the change in plasma concentration of hepcidin (ng/ml) from baseline to 6 months in participants with Gaucher disease type 1

SECONDARY OUTCOMES:
Change in Blood Glutathione Concentration | 6 months
  Outcome will be reported as the change in blood concentration of glutathione (umol/g) from baseline to 6 months in participants with Gaucher disease type 1
Change in Plasma Tumor Necrosis Factor (TNF)-alpha Concentration | 6 months
  Outcome will be reported as the change in blood concentration of TNF-alpha (pg/ml) from baseline to 6 months in participants with Gaucher disease type 1

CONTACTS AND LOCATIONS:
Overall Officials: Reena Kartha, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States